CLINICAL TRIAL: NCT04034290
Title: A Double-blind Randomized Placebo-controlled Study of Safety and Immunogenicity of Medicinal Product With a Period of Open Safety Assessment in Two Modes of Administration, in Healthy Volunteers
Brief Title: A Double-blind Randomized Placebo-controlled Study Study of the Safety, Reactogenicity and Immunogenicity of the GamFluVac
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gamaleya Research Institute of Epidemiology and Microbiology, Health Ministry of the Russian Federation (Other)
Collaborators: Main military clinical hospital named after academician N. N. Burdenko (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 03 - GamFluVac-2019
Record Dates: First submitted 2019-07-24; First posted 2019-07-26 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: influenza; vaccine; Immunologic Factors; Respiratory Tract Infections; vector vaccines
MeSH Terms: conditions — Influenza, Human; Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: This clinical trial on the second stage is designed as a double blind randomized placebo-controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Stage 1 (GamFluVac intranasal drip) (Experimental): The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) × 1011 VP/dose administrated by intranasal drip
  Interventions: Biological: GamFluVac
- Stage 1 (GamFluVac with the help of a spray dispenser) (Experimental): The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) × 1011 VP/dose administrated intranasally with the help of a spray dispenser
  Interventions: Biological: GamFluVac
- Stage 2 Vaccine (Experimental): The total number of recombinant pseudo-adenoviral particles (2.5 ± 1.25) × 1011 VP/dose
  Interventions: Biological: GamFluVac
- Stage 2 (Controll Group) (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: GamFluVac — The drug is a vaccine that induces high-level immunity against influenza A viruses
  Arms: Stage 1 (GamFluVac intranasal drip); Stage 1 (GamFluVac with the help of a spray dispenser); Stage 2 Vaccine
Other: Placebo — Placebo
  Arms: Stage 2 (Controll Group)

SUMMARY:
The aim of the present study is at the first stage: a comparative assessment of the safety of the two methods of vaccine administration, at the second - an assessment of the safety and state of post-vaccination immunity at different times after vaccination

DETAILED DESCRIPTION:
In the first stage estimate of safety of vaccine after its single administration to the nasal cavity by the drip method or by spray - dispenser during the period of observation in 30 days with the participation of 24 volunteers, divided into 2 groups of 12 people for each method of administration

After interim analysis of safety data is subject to the consent of the local ethics Committee of the Research Centre about the possibility of further studies of the drug - will be started the second phase of the study, which, along with continued security research, provides the definition of the parameters of immunogenicity of the study drug. The second phase of the study will included 200 participants, including 100 people will receive the study drug and 100 will be a control group of observation - that is, will get a placebo.

ELIGIBILITY:
Inclusion Criteria

* Men and women aged 18 to 55 years old.
* Written informed consent.
* consent to the use of effective contraceptive methods throughout the study period *

  * using one of the following methods: abstinence, condoms (male or female with or without spermicide), diaphragm or cervical cap with spermicide, intrauterine device
* body mass index (BMI) from 18.5 to 30.
* absence of acute infectious diseases or exacerbation of chronic infections at the time of vaccination and 7 days before vaccination;
* absence of allergic diseases of a serious degree (anaphylactic shock, Quincke's edema, polymorphic exudative eczema, serum sickness)
* absence of strong post-vaccination reactions or post-vaccination complications for previous use of immunobiological drugs;
* absence of pathology from the gastrointestinal tract, liver, kidneys, cardiovascular system, central nervous system, musculoskeletal system, genitourinary and endocrine systems, which may influence the evaluation of the results of the study, in the anamnesis and also according to the screening examination data;
* negative pregnancy test (for fertile women);
* negative tests for HIV, hepatitis B and C, syphilis;
* negative urine test for traces of drugs;
* negative test for alcohol content in the exhaled air;
* absence of malignant blood diseases;
* absence of malignant neoplasms;
* indicators of the total blood test at the screening not higher/lower than 1.1 x LLN/ULN (upper/lower limit of the normal reference range) *;

  * normal reference values of the laboratory performing the studies must be provided before the volunteer screening begins
* according to the biochemical blood test at the screening: the level of urea, creatinine, alanine aminotransferase, aspartate aminotransferase, glucose, creatine phosphokinase, total protein, bilirubin, glucose, LDH, alkaline phosphatase, LDL / HDL / VLDL - no higher/lower 1.1 X LLN/ULN (upper/lower limit of the normal reference range), total cholesterol level from 3,6 mmol/l to 7,8 mmol/l;
* no changes in myocardium of inflammatory or dystrophic nature according to ECG results at screening;
* lack of vaccination against influenza within 6 months before the start of the study (including during participation in other clinical trials).

Exclusion criteria

* participation of a volunteer in any other study in the last 90 days;
* any vaccination in the last 30 days;
* vaccination against influenza within 6 months before the start of the study (including during participation in other clinical trials).
* symptoms of respiratory illness in the last 3 days;
* recent frequent nasal bleeding (> 5 last year);
* chronic rhinitis, the presence of defects of the nasal septum, polyps of the nose or other significant anomalies;
* surgical operations or a history of nasal trauma for 6 months.
* treatment with steroids in the last 10 days;
* administration of immunoglobulins or other blood products for the last 3 months;
* taking immunosuppressive drugs and / or immunomodulators within 6 months before the start of the study;
* regular past or current use of narcotic drugs;
* pregnancy or breastfeeding;
* systolic blood pressure less than 100 mmHg or higher than 139 mmHg; diastolic blood pressure less than 60 mmHg. or above 90 mmHg; the heart rate is less than 60 beats per minute or more than 90 beats per minute;
* exacerbation of allergic diseases, the presence of anaphylactic reactions or angioedema in medical history;
* hypersensitivity or allergic reactions to the administration of any vaccine in medical history;
* allergic reactions to vaccine components;
* diabetes mellitus or other forms of impaired glucose tolerance;
* the presence of a concomitant disease that may influence the evaluation of the results of the study: active forms of tuberculosis, chronic liver and kidney diseases, severe thyroid dysfunction and other endocrine system diseases (diabetes mellitus), severe deseases of hematopoietic system, epilepsy and other CNS diseases, myocardial infarction, myocarditis, endocarditis, pericarditis, coronary heart disease, autoimmune pathology, serious chronic diseases requiring a hospitalisation;
* donor blood donation (450 ml and more blood or plasma) less than 2 months before the start of the study;
* taking a history of more than 5 units of alcohol (equal 0.25 liters of ethanol) per week;
* smoking: more than 10 cigarettes a day;
* planned hospitalization and / or surgical intervention during the study period, and 4 weeks before the expected date of vaccination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 224 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events | through the whole study, an average of 180 days
  Determination of Number of Participants With Adverse Events
Antibody levels a measured by an enzyme-linked immunosorbent assay (ELISA) | through the whole study, an average of 90 days
  Determination of antibody levels measured by an ELISA vs. baseline values and vs placebo

SECONDARY OUTCOMES:
Assessment of antigen-specific cell-mediated immune response | at days 0 and 7
  determination of specific T-cell- mediated response vs. baseline values ans vs placebo

CONTACTS AND LOCATIONS:
Overall Officials: Irina Gagarina, MD, PhD, Principal Investigator — Federal state budgetary institution " Main military clinical hospital named after academician N. N. Burdenko " of the Ministry of Defence of the Russian Federation
Locations (1):
- Federal state budgetary institution " Main military clinical hospital named after academician N. N. Burdenko " of the Ministry of Defence of the Russian Federation, Moscow, Russia

IPD SHARING:
Plan to Share IPD: No